CLINICAL TRIAL: NCT06428435
Title: Next Generation Home Vision Assessment
Acronym: NGHVA
Status: Completed | Type: Observational
Sponsor: NHS Forth Valley (Other Government)
Collaborators: Birmingham Children's Hospital (Other); NHS Fife (Other Government); NHS Highland (Other)
Responsible Party: Sponsor
Other Study IDs: FV1275; 286078 (Other: IRAS Project ID); 20/WM/0285 (Other: REC Number); 136640 (Other: Edge ID)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Amblyopia; Vision; Low, One Eye (Other Eye Normal); Pediatric Disorder
Keywords: teleophthalmology; remote consultations; amblyopia; paediatrics; telemedicine; digital health
MeSH Terms: conditions — Amblyopia | interventions — Vision Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ibis: Tested with Ibis technology
  Interventions: Diagnostic Test: Vision Test
- Optonet: Tested with Optonet Technology
  Interventions: Diagnostic Test: Vision Test

INTERVENTIONS:
Diagnostic Test: Vision Test — Remote vision testing via digital screen

SUMMARY:
Comparison of live remote paediatric digital vision testing outcomes versus face to face appointments in orthoptic clinic

DETAILED DESCRIPTION:
Study Overview The "Next Generation Home Vision Assessment" study aims to evaluate the feasibility and accuracy of conducting vision assessments at home using a web-based platform. This prospective, non-interventional, multi-center study will compare home-based vision tests with traditional hospital-based assessments.

Study Background The COVID-19 pandemic has significantly limited patients' ability to attend in-person eye clinic appointments, impacting vision assessments and management. Ramifications in delays continue to have an impact.

Study Rationale This study seeks to validate home-based vision assessments against standard in-person evaluations to ensure patients can be effectively monitored and managed remotely. The use of a web-based platform for vision tests could offer a reliable alternative, reducing hospital visits and maintaining care standards.

Objectives and Endpoints Primary Objective: To compare the accuracy of home-based visual acuity tests to hospital-based assessments.

Secondary Objectives: To evaluate other aspects of visual function (e.g., visual fields, color vision, contrast sensitivity) and measure patient engagement and test duration.

Study Design Type: Prospective, non-interventional Participants: Adults and children attending hospital eye services Sample Size: 360 completed assessments Duration: Minimum of 6 months

Study Procedure Participants attending hospital eye services will be recruited and provided with a patient information leaflet. Those willing to participate will undergo a visual acuity test +/- additional vision tests (secondary outcomes) during a video consultation. Hospital-based assessment results will be compared to home-based test results to determine accuracy.

ELIGIBILITY:
Inclusion criteria

- Patients attending hospital eye services will be eligible for enrolment.

Age: less than 90 years old English speakers, as no available resource for translation services. Parents / patients must be able to provide consent Patient must be able to communicate what he / she sees on a vision assessment chart.

Must have access to smartphone, tablet or home computer that can run video conferencing platforms.

Exclusion criteria

Non English speakers or lack of ability to consent Inability to communicate what is seen on a chart, or inability to complete a preferential looking visual acuity test Inability to connect to a video conferencing platform.

Ages: 0 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending hospital and at home
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Acuity | 2 weeks
  Home versus Remote Acuity difference

SECONDARY OUTCOMES:
Colour Vision | 2 weeks
  Digital versus in clinic standard
Visual field | 2 weeks
  Digital versus in clinic standard

CONTACTS AND LOCATIONS:
Overall Officials: Iain Livingstone, MBChB MD, Principal Investigator — NHS Forth Valley
Locations (4):
- United Kingdom (4):
  - Birmingham Womens and Childens Hospital, Birmingham, Birmingham
  - NHS Fife, Inverness, Inverness
  - NHS Forth Valley Research & Development Office, Falkirk, Stirlingshire
  - NHS Greater Glasgow & Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available as part of publication
Time Frame: Aim: 12 months post completion of study
Access Criteria: Open Access